CLINICAL TRIAL: NCT02654964
Title: A Phase 0/1 Study of Combination Drug Therapy For Glioblastoma Based on Personalized Cancer Stem Cell (CSC) High-Throughput Drug Screening (HTS)
Brief Title: Cancer Stem Cell High-Throughput Drug Screening Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTS Drug Screening Study
Record Dates: First submitted 2015-11-19; First posted 2016-01-13 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Drug Therapy, Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): A Drug Combination Treatment will be determined through High Throughput Screening. The classes of drugs this combination therapy will be comprised from are:
  Antineoplastic Anti-infective Antiemetic Antihyperlipidemic Anti-inflammatory Antihistamine Antihypertensive Antidepressant Cardiotonic Alcohol antagonist Diuretic Antipsychotic NMDA receptor antagonist Antidiabetic Immunosuppressant Anticonvulsant Antimethemoglobinemic Sclerosing agent
  Interventions: Drug: Combination Drug Therapy

INTERVENTIONS:
Drug: Combination Drug Therapy — Up to 3 of 73 possible interventions from the drug classes listed below will be selected based on their potency against CSCs, potential for synergy without cross-reactive toxicities, drug safety profiles, pharmacokinetics, and drug-drug interactions. Those patients that have GBM that has recurred (as defined by RANO (45)), and for whom HTS was successfully completed, will be eligible to continue to the treatment component of the study to receive the drug cocktail comprised from the following drug classes:
  Antineoplastic Anti-infective Antiemetic Antihyperlipidemic Anti-inflammatory Antihistamine Antihypertensive Antidepressant Cardiotonic Alcohol antagonist Diuretic Antipsychotic NMDA receptor antagonist Antidiabetic Immunosuppressant Anticonvulsant Antimethemoglobinemic Sclerosing agent

SUMMARY:
A study to determine the safety of CSC/ HTS-based combination drug therapy in subjects who have GBM that has recurred or progressed following prior radiation therapy and TMZ.

DETAILED DESCRIPTION:
This protocol describes a prospective single-center Phase 0/1 open-label study to evaluate the safety and efficacy of a high-throughput drug sensitivity assay to predict targeted therapies for patients who have GBM that has recurred or progressed following prior radiation therapy and TMZ. The underlying hypothesis is that treatment of patients with up to 3 lead candidates identified from individualized CSC/ HTS assays will safely (1) delay disease progression, and (2) increase survival. There is an abundance of literature strongly supporting the importance of a regimen for targeting CSCs and preventing tumor recurrence, as an additional strategy to improve the overall prognosis of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Determined at pre-screening:

* A histological diagnosis of GBM [WHO grade IV].
* Subjects ≥18 years of age
* Signed informed consent for tumor collection prior to initiation of any study-specific procedure. The patient or the patient's legal authorized representative must be able to provide written informed consent (ICF) and understand the potential risks and benefits from study enrollment and treatment
* Patients must have a life expectancy of >12 weeks

Determined at or around surgery, and prior to performing HTS:

* Patients must have a surgically accessible tumor with the intent for a gross or near total resection of the tumor mass (GBM, WHO grade IV)
* Collection of sufficient tumor material for processing CSCs

Determined at or around tumor recurrence, and after completion of HTS:

• Disease progression following radiation and TMZ therapy (as defined by RANO criteria (45); Appendix 3). Unlimited relapses are allowed, provided the functional status and other eligibility criteria for enrollment are met

Determined at baseline:

* Signed informed consent for CSC/HTS based therapy prior to initiation of any study-specific procedure or treatment. The patient or the patient's legal authorized representative must be able to provide written informed consent (ICF) and understand the potential risks and benefits from study enrollment and treatment
* Patients must have a KPS rating of ≥70 (see Appendix 4: Karnofsky Performance Scale)
* Patients must have recovered from the toxic effects of prior therapy to < Grade 2 toxicity per NCI CTCAE version 4 (Appendix 6) prior to Day 1 of Cycle 1. The minimum duration required between prior therapy and initiation of study drug treatment is as follows:

  * At least 12 weeks from completion of radiation therapy except if there is unequivocal evidence for tumor recurrence (such as histological confirmation) in which case at least 4 weeks from completion of radiation will suffice
  * 4 weeks from prior cytotoxic chemotherapy
  * 4 weeks from prior experimental drug
  * 6 weeks from nitrosoureas
  * 3 weeks from procarbazine
  * 1 week for non-cytotoxic agents.
* Subjects must have adequate renal, hepatic and bone marrow function based on screening laboratory assessments. Baseline hematologic studies and chemistry and coagulation profiles must meet the following criteria:
* Hemoglobin (Hgb)> 8 g/dL
* Absolute Neutrophil Count (ANC) > 1,000/mm3
* Platelet count > 100,000/mm3
* Creatinine < 2 mg/dL
* Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) < 3x upper limit of normal (ULN)
* Patients of childbearing potential must agree to use an adequate method of contraception for the duration of the study, and for 90 days following discontinuation of study drugs
* Females of childbearing potential must have a negative pregnancy test
* Patients must be negative for HIV, Hepatitis B and C
* Patients are cooperative and able to complete all the assessment procedures.

Exclusion Criteria:

* Any condition, including the presence of clinically significant laboratory abnormalities, which places the subject at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study
* Active infection, (including known Acquired Immunodeficiency Syndrome (AIDS) and Hepatitis C) within 3 days prior to the study enrollment
* Diseases or conditions that obscure toxicity or dangerously alter drug metabolism
* Serious intercurrent medical illness (e.g., symptomatic congestive heart failure)
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from providing informed consent unless they have a legal authorized representative that can consent on their behalf
* Inadequately controlled hypertension (defined as systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months
* History of stroke or transient ischemic attack within 6 months
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months
* History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Grade 2 or higher peripheral neuropathy per NCI CTCAE version 4
* History of abdominal fistula or gastrointestinal (GI) perforation within 6 months.
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Allergies to reagents used in this study
* Women of child bearing age not willing to use a reliable form of contraception
* Pregnancy (positive pregnancy test) or lactation
* Patient is positive for HIV, Hepatitis B or C
* Concurrent use of enzyme-inducing anti-epileptic drugs (EIAEDs) Patients must discontinue an EIAED at least two weeks prior to starting study drug
* Concurrent use of herbal medications
* Patient is simultaneously participating in another clinical trial during the Phase 1 (treatment phase) of this study. Patients may enroll/consent in the Phase 0 portion of this study for tissue collection and HTS while being treated with standard of care or clinical trial for newly diagnosed GBM prior to recurrence. Inability or unwilling to comply with protocol or study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Tumor size | 1 year
Progression free survival | 1 year
Overall response rate | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cobbs, MD, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States